CLINICAL TRIAL: NCT06953050
Title: SELF-CARE IN PARKINSON'S DISEASE: A STUDY ON PATIENTS AND CAREGIVERS/Self-care in the Patient-caregiver Dyad With Parkinson's Disease: A Descriptive Observational Study
Acronym: SPES
Status: Not yet recruiting | Type: Observational
Sponsor: Giovanni Muttillo (Other)
Responsible Party: Sponsor-Investigator, Giovanni Muttillo, Director of Nursing Services Giovanni Muttillo, ASST Gaetano Pini-CTO
Organization: ASST Gaetano Pini-CTO (Other)
Other Study IDs: ID 5732 parere numero 5732_12
Record Dates: First submitted 2025-04-22; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease (PD); Self-Care Ability
Keywords: malattia di parkinson; self-care; nurse
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patient
- Group 2: Caregiver

SUMMARY:
This descriptive observational study will involve dyads of Parkinson Disease patients and their caregivers. Participants will be recruited from the Parkinson's Disease and Movement Disorders Centre of ASST Gaetano Pini-CTO. Validated questionnaires, such as the WHOQOL-Bref, the Self-care of Chronic Illness Inventory version 2, and the Caregiver Self-efficacy in Contributing to Self-care Scale, will be administered. The study will also include semi-structured interviews to gather qualitative data on the patients' and caregivers' perceptions of self-care. A non-probabilistic convenience sampling method will be used, with the inclusion of both patients at any disease stage and their primary caregivers. The sample size will range 311 dyads with 5% margin of error.

DETAILED DESCRIPTION:
The primary objective of this study is to describe the proportion of self-care maintenance in the population with Parkinson's Disease and their respective caregivers. Gaining an in-depth understanding of the phenomenon in its experiential and perceptual components, as well as the meanings attributed to it, is essential for developing and validating a new tool capable of assessing and measuring self-care in Parkinson's Disease. The secondary objectives are (a) to describe the proportions of self-care monitoring and management in the population with Parkinson's Disease and their respective caregivers; (b) to explore the meaning attributed by patients with Parkinson's Disease to self-care in its three dimensions: self-care maintenance, monitoring, and management; (c) to describe the attitudes and self-care behaviours adopted by patients with Parkinson's Disease across different disease stages; (d) to explore the meaning attributed by caregivers of patients with Parkinson's Disease to self-care in its three dimensions: self-care maintenance, monitoring, and management; (e) to describe the attitudes and self-care behaviours adopted by caregivers of patients with Parkinson's Disease across different disease stages; (f) to identify the dimensions of self-care and the constructs that should be represented within the items of the new instrument, the Parkinson's Disease Self-care Questionnaire (PDSC-Q).

ELIGIBILITY:
Inclusion Criteria:

* Spatial-temporal orientation
* Identifying as the primary caregiver of the person
* Understanding of the Italian language
* Consent to participate in the study
* Informal caregiver

Exclusion Criteria:

* Secondary forms of Parkinson's Disease
* Subjects with cognitive impairments, assessed with the Mini Mental State Examination; score lower than 24/30 Subjects who do not understand written and spoken Italian Subjects who did not provide consent to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Caregivers and patients with idiopathic Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 311 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Self-care | Baseline
  Self Care of Chronic Illness Inventory versione 2
Self-care caregiver | Baseline
  Caregiver Self-efficacy in Contributing to self-care scale (CSE-CSC)

SECONDARY OUTCOMES:
Perception of quality of life | Baseline
  WHOQOL-BREF

IPD SHARING:
Plan to Share IPD: No
SHARING WITH OTHER RESEARCHERS IS NOT NECESSARY

REFERENCES:
- [Derived] Petralito M, Tedesco C, Isaias IU, Muttillo G, Castaldo A, Pucciarelli G, Caruso R. Self-care and its assessment in the patient-caregiver dyad in Parkinson's disease: a mixed-method study protocol. BMJ Open. 2025 Nov 4;15(11):e107471. doi: 10.1136/bmjopen-2025-107471. PMID 41193192